CLINICAL TRIAL: NCT06271577
Title: Smartphone Twelve-Lead ECG Utility In ST-Elevation Myocardial Infarction II (STLEUISII)
Brief Title: Smartphone Twelve-Lead ECG Utility In ST-Elevation Myocardial Infarction II
Acronym: STLEUISII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AliveCor (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO-0013
Record Dates: First submitted 2024-02-12; First posted 2024-02-22 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Myocardial Infarction; Ischemia; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Heart Attack; Heart Failure
MeSH Terms: conditions — Myocardial Infarction; Ischemia; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- AliveCor 12-lead ECG (Experimental): A single research-related procedure will be required (i.e., an AliveCor 12-lead ECG). Effort will be made to ensure that the performance of this procedure will not delay any treatment and/or diagnostic procedures that are part of usual or specialized care that the patient requires.
  Interventions: Device: AliveCor 12-lead ECG

INTERVENTIONS:
Device: AliveCor 12-lead ECG — The primary objective of this study is to determine if the AliveCor 12-lead Smartphone ECG is an acceptable substitute for a standard 12-lead ECG in the identification of STEMI and NSTEMI.

SUMMARY:
AliveCor (www.alivecor.com) has developed several electrocardiogram (ECG) devices that interface with iOS and Android smartphones and tablets via various Kardia apps. The current Kardia family of devices can measure single lead and six limb-lead ECGs, depending on the device. KardiaMobile, KardiaMobile 6L, and KardiaMobile Card have FDA clearance for ECG rhythm recording. A modified single-lead Kardia smartphone 12-lead ECG was previously validated in the multicenter ST LEUIS study for the diagnosis of ST-Segment Elevation Myocardial Infarction (STEMI) and Non-ST-Elevation Myocardial Infarction (NSTEMI).

Recently, AliveCor developed a new device: AliveCor (AC) 12-lead (12L) ECG System to record simultaneously 4 leads of ECG and then generate complete 12-lead ECGs. A previous protocol at the University of Oklahoma involved 200 subjects with early prototypes of the AC 12L device with the specific aim to validate that it accurately generated 12-lead ECGs as compared to simultaneously acquired FDA-cleared 12-lead ECGs. The prototype version of the AliveCor 12L ECG System simultaneously measured four channels of ECG (leads I, II, V2, V4), calculated the remaining limb leads as is standard for 12-lead ECGs (Leads III, aVR, aVL, aVF) and synthesized the remaining 4 precordial ECG leads (V1, V3, V5, V6). This protocol will serve to validate the production version of the system against standard 12-Lead ECGs for the diagnosis of STEMI and NSTEMI in patients admitted to the Emergency Department or directly to the Cardiac Cath Lab for the evaluation of chest pain. It is anticipated that the waveforms for each of the 12 leads from the AC 12L ECG System will be highly correlated with the corresponding leads from the comparator commercially available 12-lead ECG devices used at participating sites. The purpose of this study is to clinically validate that the four-channel AC 12L ECG device can enable the diagnosis of STEMI and NSTEMI in a non-inferior manner to existing 12-lead ECG devices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years of age.
* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.
* Symptoms of chest pain upon presentation at the Emergency Department of the participating institution.

Exclusion Criteria:

* Inability or refusal of the patient and/or the patient's legally acceptable representative to provide written informed consent for any reason.
* Other conditions that in the opinion of the Lead Investigator may increase risk to the subject and/or compromise the quality of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Inter-rater variability for Standard 12-lead ECG readings | 30 seconds
Inter-rater variability for AC 12L ECG readings | 30 seconds
Number of standard 12-lead ECG readings requiring a consensus consultation | 30 seconds
Number of AC 12L ECG readings requiring a consensus consultation | 30 seconds
Sensitivity of AC 12L ECGs requiring consensus consultation, compared to standard 12-lead ECG requiring consensus consultation, for the diagnosis of STEMI | 30 seconds
Specificity of AC 12L ECGs requiring consensus consultation, compared to standard 12-lead ECG requiring consensus consultation, for the diagnosis of STEMI | 30 seconds
Positive predictive value of AC 12L ECGs requiring consensus consultation, compared to standard 12-lead ECG requiring consensus consultation, for the diagnosis of STEMI | 30 seconds
Negative predictive power of the AC 12L ECGs requiring consensus consultation, compared to standard 12-lead ECG requiring consensus consultation, for the diagnosis of STEMI | 30 seconds
Mean subjective correlation score for AC 12L ECGs in which the standard 12-lead ECG diagnosis is STEMI | 30 seconds
Mean subjective correlation score for AC 12L ECGs in which the standard 12-lead ECG diagnosis is not STEMI | 30 seconds
Mean summative ST-segment elevation, summative ST-segment depression and summative ST-segment deviation for AC 12L ECGs compared to standard 12-lead ECGs | 30 seconds

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Intermountain Health, Murray, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muhlestein JB, Anderson JL, Bethea CF, Severance HW, Mentz RJ, Barsness GW, Barbagelata A, Albert D, Le VT, Bunch TJ, Yanowitz F, May HT, Chisum B, Ronnow BS, Muhlestein JB; Duke University Cooperative Cardiovascular Society (DUCCS) investigators. Feasibility of combining serial smartphone single-lead electrocardiograms for the diagnosis of ST-elevation myocardial infarction. Am Heart J. 2020 Mar;221:125-135. doi: 10.1016/j.ahj.2019.12.016. Epub 2019 Dec 27. PMID 31986289